CLINICAL TRIAL: NCT04792918
Title: Intestinal Microbiome Strain-level Stability in NEC/ or LOS Patients
Brief Title: Characterization of Intestinal Microbiota Stability in Preterm Born Neonates
Acronym: NEC
Status: Completed | Type: Observational
Sponsor: Emma Marie Caroline Slack (Other)
Collaborators: University of Zurich (Other); University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor-Investigator, Emma Marie Caroline Slack, Prof. Dr., ETH Zurich
Organization: ETH Zurich (Other)
Other Study IDs: NEC
Record Dates: First submitted 2021-03-09; First posted 2021-03-11 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Necrotising Enterocolitis; Late-Onset Neonatal Sepsis
MeSH Terms: conditions — Enterocolitis, Necrotizing; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NEC/LOS preterm infants: Collection of biological samples (stool, stomach fluid, blood) and health-related data over the first few weeks of life, additional stool samples after onset of NEC/LOS
- Preterm infants not developing NEC/LOS: Collection of biological samples (stool, stomach fluid, blood) and health-related data over the first few weeks of life
- Family members of preterm infants: Collection of biological samples (stool, breastmilk, vaginal swab) and health-related data at one timepoint after the birth of the preterm infant from members of the family (mother, father)

SUMMARY:
Study around very-low birthweight preterm infants at high risk of developing necrotizing enterocolitis (NEC) or late-onset sepsis (LOS). Collection of stool and other biological samples to assess the strain-level stability of gastrointestinal microbiota in these preterm infants who may or may not develop NEC/LOS.

DETAILED DESCRIPTION:
This study aims to collect biological samples (stool, stomach fluid, and blood) from preterm infants at risk of developing NEC or LOS; as well as environmental samples from infants' hospital surroundings (swabs, air), nutritional intake (formula, breastmilk) and samples from their family members (faeces, vaginal swab).

The main focus of the study is to assess strain-level stability of gastrointestinal microbiota in these infants and potentially assess the source of disease-causing microbiota species/strains.

ELIGIBILITY:
Inclusion Criteria:

-Preterm infants with a gestational age < 32 weeks or a birthweight < 1500g and their family members

Exclusion Criteria:

* Intestinal atresia
* Live born infants referred to from other hospitals later than 3 days after birth

Ages: 0 Days to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population is represented by infants born at gestational age below 32 weeks (very preterm born infants) or with a birthweight below 1500g (very low birthweight infants). It is estimated that approximately 100 infants will be enrolled during the study period. As the aim is to study stability of the premature microbiota within individual patients, the study design precludes the need of control groups.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Strain-level stability | 24 months
  Identify members of the gastrointestinal microbiota (species/strains) that are associated with development of NEC or LOS in very-low birthweight/very preterm Identify members of the gastrointestinal microbiota (species/strains) that are associated with development of NEC or LOS in very-low birthweight/very preterm infants via changes in frequencies, absolute colonization levels, or temporal stability

SECONDARY OUTCOMES:
Source of bacterial species/strains | 24 months
  Quantify genetic similarity between potentially disease-causing microbiota strains found within NEC/LOS patients and within family members (faeces, breastmilk, vaginal swab) and hospital surroundings

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Children's Hospital Zürich, Zurich
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No